CLINICAL TRIAL: NCT04699500
Title: Spanish Validation and Cross-cultural Adaptation of the QoR-15 Post-anesthetic Recovery Quality Questionnaire: The QoR-15E
Brief Title: Spanish Validation and Cross-cultural Adaptation of the QoR-15E
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)620/2020
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Humans; Reproducibility of Results; Cross-Cultural Comparison; Surveys and Questionnaires; Postoperative Period; Anesthetics; Perception
Keywords: Quality; Recovery; Anesthesia; Validation; Adaptation; Spanish

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The satisfactory recovery of the patient after a surgery with an anesthetic request is very important for a quality and excellence assistance. The quality of recovery questionnaire QoR-15 was validated by their authors in 2013 with the study titled development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. This questionnaire allows a comprehensive assessment by associating the physiological parameters until then assessed with the subjective personal perception of the patient of his state of health. With the consent of its original author, this study is carried out to validate the questionnaire in Spanish and adapted to our environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Comprehensive and sign informed consent.
* Knows and understands the Spanish language.
* Undergo a scheduled surgical intervention under any type of anesthetic procedure from the specialties of general surgery, urology and gynecology.
* Score > 26 points in the Mini Mental State Examination (MMSE) test.

Exclusion Criteria:

* Patients under 18 years old.
* Not having signed the informed consent.
* Not knowing or understanding the Spanish language.
* Surgical intervention from other specialties than general surgery, urology and gynecology.
* Score < 27 points in the Mini Mental State Examination (MMSE) test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population will be made up of adult patients who undergo a surgical intervention as a therapeutic or diagnostic procedure (general surgery, urology and gynecology) that require an anesthetic technique in the General Area of the Vall d'Hebron University Hospital, whose intended destination after the procedure would be the post-anesthetic recovery unit, before hospital discharge
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Spanish version of the Quality of Recovery 15 questionnaire: The QoR-15E. | 1 year
  The aim of this study is to carry out cross-cultural adaptation and validate the postoperative questionnaire QoR-15 to the Spanish environment and evaluate its validity and reliability.
  This questionnaire consists of 15 items with a total score of 150 points where 150 points is better than 0 points for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Manrique Muñoz, MD, PhD, Study Director — Hospital Vall d'Hebron; Miriam de Nadal Clanchet, MD, PhD, Study Director — Hospital Vall d'Hebron
Locations (1):
- Comitè Ètic d'Investigació Clínica HUVH, Barcelona, Spain

REFERENCES:
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Kleif J, Edwards HM, Sort R, Vilandt J, Gogenur I. Translation and validation of the Danish version of the postoperative quality of recovery score QoR-15. Acta Anaesthesiol Scand. 2015 Aug;59(7):912-20. doi: 10.1111/aas.12525. Epub 2015 Apr 13. PMID 25867135
- [Background] Sa AC, Sousa G, Santos A, Santos C, Abelha FJ. Quality of Recovery after Anesthesia: Validation of the Portuguese Version of the 'Quality of Recovery 15' Questionnaire. Acta Med Port. 2015 Sep-Oct;28(5):567-74. doi: 10.20344/amp.6129. Epub 2015 Oct 30. PMID 26667859
- [Background] Llamas-Velasco S, Llorente-Ayuso L, Contador I, Bermejo-Pareja F. [Spanish versions of the Minimental State Examination (MMSE). Questions for their use in clinical practice]. Rev Neurol. 2015 Oct 16;61(8):363-71. Spanish. PMID 26461130
- [Background] Demumieux F, Ludes PO, Diemunsch P, Bennett-Guerrero E, Lujic M, Lefebvre F, Noll E. Validation of the translated Quality of Recovery-15 questionnaire in a French-speaking population. Br J Anaesth. 2020 Jun;124(6):761-767. doi: 10.1016/j.bja.2020.03.011. Epub 2020 Apr 15. PMID 32303379